CLINICAL TRIAL: NCT02088424
Title: Insulin Resistance and Recurrent Abortion
Brief Title: the Insulin Resistance in Recurrent Miscarriage IN RECURRENT ABORTION
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohamed ahmed selem, THE ROLE OF INSULIN RESISTANCE IN RECURRENT MISCARRIAGE, Ain Shams University
Other Study IDs: mohd-1978
Record Dates: First submitted 2014-03-08; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Recurrent Abortion
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group A: cases with recurrent abortion with insulin resisance
  Interventions: Other: insulin resistance(fasting glucose/fasting insulin)
- GROUP B: cases that are pregnant with no history of recurrent abortion with no insulin resistance
  Interventions: Other: insulin resistance(fasting glucose/fasting insulin)

INTERVENTIONS:
Other: insulin resistance(fasting glucose/fasting insulin) — insulin resistance(fasting glucose/fasting insulin )

SUMMARY:
THE INSULIN RESISTANCE IN RECURRENT ABORTION

DETAILED DESCRIPTION:
THE ROLE OF INSULIN RESISTANCE IN RECURRENT ABORTION

ELIGIBILITY:
Inclusion Criteria:

1. Women in the child bearing period between 23-40 years.
2. All patients are pregnant.
3. The gestational age of both groups 6-13 weeks

Exclusion Criteria:

1. Patients with gestational diabetes and gestational impaired glucose tolerance.
2. The patients who took medication that could affect glucose metabolism at the time of the study
3. Patients with other causes of recurrent abortion as(thyroid dysfunction, uterine anomalies chromosomal abnormalities, antiphspholipid antibody syndrome, uterine anomalies and TORCH syndrome).
4. Patients with PCOS.
5. Obese patients(BMI>30)

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Women in the child bearing period between 23-40 years.
  2. All patients are pregnant.
  3. The gestational age of both groups 6-13 weeks
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-11 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose | 3 month
  Click here for more information about this study: the role of insulin resistance in recurrent abortion

SECONDARY OUTCOMES:
fasting Insulin | 3 month

OTHER OUTCOMES:
oral glucose tolerance test | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams maternity hospital, Cairo, Egypt